CLINICAL TRIAL: NCT06640309
Title: The Effect of Nicotinamide on the Clinical Outcome of Rheumatoid Arthritis Patients
Acronym: NAM&RA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara ahmed raslan, clinical pharmacist at Ain Shams University Hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAM/RA/1223
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Nicotinamide; Quality of life; DAS-28
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled interventional parallel open label study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide group (Experimental): Patients will receive nicotinamide 1000mg tablet once daily.in addition to their conventional therapy for three months.
  Interventions: Drug: Nicotinamide Tablet; Drug: conventional synthetic antirheumatic drugs
- control group (Active Comparator): Patients will receive their conventional therapy only.
  Interventions: Drug: conventional synthetic antirheumatic drugs

INTERVENTIONS:
Drug: Nicotinamide Tablet — Nicotinamide is anti-inflammatory and antioxidant.
  Arms: Nicotinamide group
Drug: conventional synthetic antirheumatic drugs — methotrexate- leflunomide- sulfasalazine- hydroxychloroquine

SUMMARY:
A randomized controlled interventional study to evaluate the efficacy and safety of nicotinamide supplementation in rheumatoid arthritis patients receiving conventional synthetic disease modifying anti-rheumatic drugs.

DETAILED DESCRIPTION:
Study design:

A prospective randomized controlled interventional parallel open label study.

Patient randomization:

All patients fulfilling the inclusion criteria will be randomly assigned by simple randomization into either nicotinamide group or control group as follows:

* Nicotinamide group: consists of thirty-five patients who will receive nicotinamide 1000mg tablet once daily.in addition to their conventional therapy.
* Control group: consists of thirty-five patients who will receive their conventional therapy only.

Methodology:

At baseline, the following will be obtained through patients' interview:

1. Demographic data.
2. Medical history and comorbidities.
3. The disease activity; identified through patients' physical examination and serum C-Reactive Protein (CRP) levels as prerequisites for Disease Activity Score-28 (DAS-28-CRP).
4. The disease duration.
5. Current medications history.

Evaluation of the efficacy and safety of nicotinamide will be assessed at baseline and after three months through:

1. Blood sampling will be collected from patients for serum CRP , Erythrocyte sedimentation rate (ESR) and analysis of Interleukin-10 .These samples will be directly centrifuged at 1000 x g for fifteen minutes and then plasma will be separated and collected in capped test tubes, then will be stored at -80 °C until analysis.

   Interleukin-10 serum level will be measured using an Enzyme Linked Immunosorbent Assay (ELISA) technique.
2. Disease Activity will be calculated based on tender joint count (TJC) and swollen joint count (SJC) following the assessment of twenty-eight joints, serum CRP level, and the patient's global health assessment (PGA) on a scale from zero to one hundred. The score will be calculated using the following equation:

   DAS-28-CRP = 0.56* √(TJC28) + 0.28* √(SJC28) + 0.36*ln (CRP + 1) +0.014*(PGA) + 0.96
3. Patient's QOL will be assessed by using the Health Assessment Questionnaire-Disability Index (HAQ-DI)
4. Patients will be educated about the side effects and/or adverse effects of nicotinamide, where, safety and tolerability will be monitored by reporting the incidence of any side effect and /or adverse effect such as stomach upset, flatulence, dizziness, headache, and rash.

Blood samples will be collected for complete blood count (CBC), alanine transaminase (ALT), aspartate transaminase (AST), serum creatinine (Scr.) levels analysis to monitor adverse effects of conventional synthetic disease-modified antirheumatic (csDMARDs) drugs and nicotinamide.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-65 years).
* Patients with a diagnosis of established rheumatoid arthritis.
* Patients presenting with moderate to high disease activity identified as disease activity score-28 based on C-reactive protein levels (DAS-28-CRP) >3.2.
* Receiving stable regimen of one or more conventional disease modifying antirheumatic drugs for at least the past three months.
* Patients willing to sign an informed consent.

Exclusion Criteria:

* Patients with a known history of hypersensitivity or drug allergies to nicotinamide
* Patients receiving nicotinamide for any other indications.
* Receiving any dosage forms/ dosage regimen of vitamin B3 supplementation
* Receiving biologic disease modified antirheumatic drugs therapy.
* Impaired liver functions (liver transaminases level ≥ three times upper normal limits).
* Impaired kidney functions (estimated glomerular filtration rate (eGFR) < 30 ml/min)
* Pregnancy and lactation.
* Patients with other auto-immune diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Disease severity assessment using DAS-28 -CRP | At baseline and after three months.
  DAS-28-CRP at baseline and at end of study, which will be calculated based on tender joint count (TJC) and swollen joint count (SJC) following the assessment of twenty-eight joints (figure 1) , serum CRP level, and the patient's global health assessment (PGA) on a scale from zero to one hundred. The score will be calculated using the following equation: (CASTREJÓN et al., 2010) DAS-28-CRP = 0.56* √(TJC28) + 0.28* √(SJC28) + 0.36*ln (CRP + 1) +0.014*(PGA) + 0.96

SECONDARY OUTCOMES:
Serum Interleukin-10 | At baseline and after three months.
  Venous blood samples will be collected from patients at baseline and at the end of the study (three months). Blood samples will be directly centrifuged at 1000 x g for fifteen minutes and then plasma will be separated and collected in capped test tubes, then will be stored at -80 °C until analysis. Interleukin-10 serum level will be measured at baseline and after three months of study period using an ELISA technique according to the manufacturer's protocol.
Detection of any change in inflammatory markers | At baseline and after three months.
  Serum C-reactive protein and Erythrocyte sedimentation rate.
Quality of Life (QOL) questionnaire | At baseline and after three months.
  Patient's QOL will be assessed by using the Health Assessment Questionnaire-Disability Index (HAQ-DI) at baseline and after three months. It assesses patient's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities
Safety and tolerability of Nicotinamide | Three months.
  Patients will be educated about the side effects and/or adverse effects of nicotinamide, where, safety and tolerability will be monitored by reporting the incidence of any side effect and /or adverse effect such as stomach upset, flatulence, dizziness, headache, and rash.

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El wakeel, Professor, Study Director — Professor and head of department of Clinical Pharmacy at Faculty of Pharmacy Ain Shams University; May Ahmed, Asst. professor, Study Director — Assistant professor of Clinical Pharmacy, Ain Shams University-Faculty of Pharmacy
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamat JP, Devasagayam TP. Nicotinamide (vitamin B3) as an effective antioxidant against oxidative damage in rat brain mitochondria. Redox Rep. 1999;4(4):179-84. doi: 10.1179/135100099101534882. PMID 10658823
- [Background] Miesel R, Kurpisz M, Kroger H. Modulation of inflammatory arthritis by inhibition of poly(ADP ribose) polymerase. Inflammation. 1995 Jun;19(3):379-87. doi: 10.1007/BF01534394. PMID 7628865
- [Background] Ungerstedt JS, Blomback M, Soderstrom T. Nicotinamide is a potent inhibitor of proinflammatory cytokines. Clin Exp Immunol. 2003 Jan;131(1):48-52. doi: 10.1046/j.1365-2249.2003.02031.x. PMID 12519385